CLINICAL TRIAL: NCT03950856
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator-controlled, Lot-to-Lot Consistency Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Healthy Adults 50 Years of Age or Older (PNEU-TRUE)
Brief Title: Lot-to-Lot Consistency of V114 in Healthy Adults (V114-020)
Acronym: PNEU-TRUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V114-020; V114-020 (Other: Merck); 2018-004266-33 (Other: EudraCT Number)
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Pneumococcal Infections; Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia, Pneumococcal | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- V114 Lot 1 (Experimental): Single intramuscular (IM) dose at 0.5 mL of V114 Lot 1 pneumococcal conjugate vaccine at Visit 1 (Day 1)
  Interventions: Drug: V114
- V114 Lot 2 (Experimental): Single IM dose at 0.5 mL of V114 Lot 2 pneumococcal conjugate vaccine at Visit 1 (Day 1)
  Interventions: Drug: V114
- V114 Lot 3 (Experimental): Single IM dose at 0.5 mL of V114 Lot 3 pneumococcal conjugate vaccine at Visit 1 (Day 1)
  Interventions: Drug: V114
- Prevnar 13™ (Active Comparator): Single IM dose at 0.5 mL of Prevnar 13™ at Visit 1 (Day 1)
  Interventions: Drug: Prevnar 13™

INTERVENTIONS:
Drug: V114 — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F in each 0.5 mL dose.
  Arms: V114 Lot 1; V114 Lot 2; V114 Lot 3
Drug: Prevnar 13™ — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F in each 0.5. mL dose.
  Arms: Prevnar 13™

SUMMARY:
The primary objectives are to evaluate the safety and tolerability of V114 and to compare the serotype-specific opsonophagocytic activity (OPA) geometric mean titers (GMTs) across 3 different lots of V114. The primary hypothesis is that all 3 lots of V114 are equivalent as measured by the serotype-specific OPA GMTs for 15 serotypes in V114 at 30 days postvaccination.

ELIGIBILITY:
Inclusion Criteria:

* Participant has good health in the opinion of the investigator. Any underlying chronic condition must be documented to be in stable condition according to the investigator's judgment.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Female participant is eligible to participate if she is not pregnant, not breastfeeding, and is not a woman of childbearing potential (WOCBP) OR a WOCBP who agrees to use agreed upon contraception during the treatment period and for at least 6 weeks after the last dose of study intervention.

Exclusion Criteria:

* History of invasive pneumococcal disease (IPD) (positive blood culture, positive cerebrospinal fluid culture, or positive culture at another sterile site) or known history of other culture-positive pneumococcal disease within 3 years of Visit 1 (Day 1).
* Known hypersensitivity to any component of pneumococcal polysaccharide vaccine, pneumococcal conjugate vaccine (PCV), or any diphtheria toxoid-containing vaccine.
* Known or suspected impairment of immunological function including, but not limited to, a history of congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or history of autoimmune disease.
* Coagulation disorder contraindicating intramuscular vaccinations.
* Recent febrile illness (defined as oral or tympanic temperature ≥100.4°F [≥38.0°C] or axillary or temporal temperature ≥99.4°F [≥37.4°C]) or received antibiotic therapy for any acute illness occurring within 72 hours before receipt of study vaccine.
* History of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* A WOCBP who has a positive urine or serum pregnancy test before the first vaccination at Visit 1 (Day 1).
* Has received any pneumococcal vaccine or is expected to receive any pneumococcal vaccine during the study outside of the protocol.
* Has received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed intervention at least 30 days before study entry.
* Has received systemic corticosteroids exceeding physiologic replacement doses (approximately 5 mg/day prednisone equivalent) within 14 days before vaccination. (Note: Topical, ophthalmic, intra-articular or soft-tissue [e.g., bursa, tendon steroid injections], and inhaled/nebulized steroids are permitted).
* Is receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease.
* Has received any non-live vaccine within the 14 days before receipt of any study vaccine or is scheduled to receive any non-live vaccine within 30 days following receipt of any study vaccine. (Exception: Inactivated influenza vaccine may be administered but must be given at least 7 days before receipt of any study vaccine or at least 15 days after receipt of any study vaccine.)
* Has received any live vaccine within 30 days before receipt of any study vaccine or is scheduled to receive any live vaccine within 30 days following receipt of any study vaccine. If this exclusion criterion is met, then Day 1 Visit may be rescheduled for a time when criterion is not met.
* Has received a blood transfusion or blood products, including immunoglobulin, within the 6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product within 30 days of receipt of study vaccine. Autologous blood transfusions are not considered an exclusion criterion.
* Currently participating in or has participated in an interventional clinical study with an investigational compound or device within 2 months of participating in this current study.
* In the opinion of the investigator, has a history of clinically relevant drug or alcohol use that would interfere with participation in protocol-specified activities.
* History or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might expose the participant to risk by participating in the study, confound the results of the study, or interfere with the participant's participation for the full duration of the study.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2340 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (55):
- United States (30):
  - Synexus Clinical Research US, Inc. ( Site 1031), Chandler, Arizona
  - Synexus ( Site 1043), Mesa, Arizona
  - Southland Clinical Research Center ( Site 1027), Fountain Valley, California
  - Valley Clinical Trials Inc. ( Site 1003), Northridge, California
  - Center for Clinical Trials, LLC ( Site 1019), Paramount, California
  - California Research Foundation ( Site 1006), San Diego, California
  - Artemis Institute for Clinical Research ( Site 1041), San Marcos, California
  - Alta California Medical Group ( Site 1020), Simi Valley, California
  - Alliance for Multispecialty Research, LLC ( Site 1029), Coral Gables, Florida
  - Accel Research Sites-DeLand Clinical Research Unit ( Site 1026), DeLand, Florida
  - Jacksonville Center for Clinical Research ( Site 1014), Jacksonville, Florida
  - L&C Professional Medical Research Institute ( Site 1012), Miami, Florida
  - Alpha Science Research ( Site 1015), Miami, Florida
  - QPS Miami Research Associates ( Site 1035), South Miami, Florida
  - Benchmark Research ( Site 1040), Metairie, Louisiana
  - Centennial Medical Group ( Site 1010), Elkridge, Maryland
  - Community Clinical Research Network (Marlboro, MA) ( Site 1025), Marlborough, Massachusetts
  - Wake Research Clinical Research Center of Nevada, LLC ( Site 1044), Las Vegas, Nevada
  - Southwest CARE Center ( Site 1011), Santa Fe, New Mexico
  - Corning Center For Clinical Research ( Site 1033), Corning, New York
  - Regional Clinical Research, Inc. ( Site 1024), Endwell, New York
  - Rochester Clinical Research, Inc. ( Site 1039), Rochester, New York
  - PMG Research of Winston Salem ( Site 1037), Winston-Salem, North Carolina
  - Unity Clinical Research ( Site 1036), Lindsay, Oklahoma
  - Coastal Carolina Research Center ( Site 1034), Mt. Pleasant, South Carolina
  - Wellness Clinical Research Associates ( Site 1038), Allen, Texas
  - Diagnostics Research Group ( Site 1042), San Antonio, Texas
  - Synexus ( Site 1000), Murray, Utah
  - Advanced Clinical Research ( Site 1028), West Jordan, Utah
  - Allegiance Research Specialists ( Site 1013), Wauwatosa, Wisconsin
- Australia (4):
  - Paratus Clinical Pty Ltd - Blacktown Clinic ( Site 6006), Blacktown, New South Wales
  - Australian Clinical Research Network ( Site 6000), Maroubra, New South Wales
  - Box Hill Hospital ( Site 6001), Box Hill, Victoria
  - Trialswest ( Site 6004), Murdoch, Western Australia
- Chile (5):
  - CESFAM Colina ( Site 2002), Santiago, RM
  - Clinica Alemana de Santiago Adolescencia ( Site 2000), Santiago, Santiago Metropolitan
  - Instituto Nacional del Torax ( Site 2004), Santiago
  - Centro de Investigacion Clinica UC CICUC ( Site 2001), Santiago
  - Hospital Dr. Hernan Henriquez Aravena ( Site 2003), Temuco
- Denmark (6):
  - Aalborg University Hospital ( Site 3003), Aalborg
  - Aarhus Universitets hospital ( Site 3004), Aarhus N
  - CCBR. Center for Clinical and Basic Research ( Site 3000), Ballerup Municipality
  - Rigshospitalet ( Site 3005), Copenhagen
  - Hvidovre Hospital ( Site 3002), Hvidovre
  - Odense Universitetshospital ( Site 3001), Odense
- Finland (7):
  - Tampereen yliopisto Etela-Helsingin Rokotetutkimusklinikka ( Site 4006), Helsinki
  - Jarvenpaan rokotetutkimuskeskus ( Site 4005), Jarvenpaa
  - Kokkolan rokotetutkimusklinikka ( Site 4002), Kokkola
  - Tampereen yliopisto Oulun rokotetutkimusklinikka ( Site 4001), Oulu
  - Tampereen yliopisto Porin rokotetutkimusklinikka ( Site 4004), Pori
  - Tampereen yliopisto - Tampereen rokotetutkimusklinikka ( Site 4000), Tampere
  - Turun rokotetutkimuskeskus ( Site 4003), Turku
- United Kingdom (3):
  - Medinova Lakeside Dedicated Research Centre ( Site 5004), Corby, Northamptonshire
  - GP Direct ( Site 5000), Harrow
  - Vauxhall Primary Health Care ( Site 5002), Liverpool

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Simon JK, Staerke NB, Hemming-Harlo M, Layle S, Dagan R, Shekar T, Pedley A, Jumes P, Tamms G, Sterling T, Musey L, Buchwald UK; V114-020 PNEU-TRUE study group. Lot-to-lot consistency, safety, tolerability, and immunogenicity of V114, a 15-valent pneumococcal conjugate vaccine, in healthy adults aged >/=50 years: A randomized phase 3 trial (PNEU-TRUE). Vaccine. 2022 Feb 23;40(9):1342-1351. doi: 10.1016/j.vaccine.2021.12.067. Epub 2022 Jan 14. PMID 35039194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy males or females ≥50 years of age without a history of invasive pneumococcal disease or prior administration of any pneumococcal vaccine were enrolled in this study.
Groups:
- Prevnar13™: Single IM dose at 0.5 mL of Prevnar 13™ at Visit 1 (Day 1)
Period: Overall Study
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Started (Randomized) | 702 | 704 | 701 | 233
Vaccinated | 698 | 704 | 700 | 231
Completed | 683 | 689 | 683 | 227
Not Completed | 19 | 15 | 18 | 6
Not completed — Death | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 5 | 6 | 8 | 2
Not completed — Protocol Violation | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 3 | 1
Not completed — Unable to phone | 7 | 6 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- V114 Lot 1: Single IM dose at 0.5 mL of V114 Lot 1 pneumococcal conjugate vaccine at Visit 1 (Day 1)
- Total: Total of all reporting groups
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™ | Total
Number analyzed (Participants) | 702 | 704 | 701 | 233 | 2340
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (7.5) | 64.4 (7.8) | 64.3 (7.4) | 64.2 (8.0) | 64.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 387 | 422 | 404 | 133 | 1346
  Male | 315 | 282 | 297 | 100 | 994
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 131 | 154 | 138 | 41 | 464
  Not Hispanic or Latino | 560 | 540 | 558 | 190 | 1848
  Unknown or Not Reported | 11 | 10 | 5 | 2 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 0 | 0 | 5
  Asian | 18 | 34 | 36 | 10 | 98
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 35 | 41 | 34 | 20 | 130
  White | 644 | 621 | 628 | 203 | 2096
  More than one race | 3 | 4 | 3 | 0 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event Following Vaccination With Separate V114 Lots
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs consisted of redness/erythema, swelling, and tenderness/pain. The 95% confidence interval (CI) were based on the exact binomial method proposed by Clopper and Pearson. Following vaccination with the three lots of V114 the percentage of participants with solicited injection-site AEs was assessed. Per the statistical analysis plan, the Prevnar 13™ treatment group was not included as it was not analyzed with the same approach as the separate V114 lots.
Time Frame: Up to Day 5
Population: Randomized participants according to the intervention they actually received. One participant randomized to the Prevnar 13™ group incorrectly received V114 Lot 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 699 | 704 | 700 | 0
Percentage of participants
  Injection site erythema | 10.2 [8.0 to 12.6] | 11.5 [9.2 to 14.1] | 11.0 [8.8 to 13.6] |
  Injection site pain | 66.1 [62.5 to 69.6] | 67.0 [63.4 to 70.5] | 67.3 [63.7 to 70.8] |
  Injection site swelling | 15.6 [13.0 to 18.5] | 15.8 [13.2 to 18.7] | 14.7 [12.2 to 17.6] |

2. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event Following Vaccination: Combined Lots of V114 or Prevnar 13™
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs consisted of redness/erythema, swelling, and tenderness/pain. Per the statistical analysis plan, within-group CIs were not calculated.
Time Frame: Up to Day 5
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- V114 Combined Lots 1,2 and 3: Single IM dose at 0.5 mL of either V114 Lots 1,2 or 3 pneumococcal conjugate vaccine at Visit 1 (Day 1)
Arm/Group | V114 Combined Lots 1,2 and 3 | Prevnar13™
Number analyzed (Participants) | 2103 | 230
Percentage of participants
  Injection site erythema | 10.9 | 9.6
  Injection site pain | 66.8 | 52.2
  Injection site swelling | 15.4 | 14.3
Statistical Analysis 1: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Injection site erythema: V114 Combined Lots - Prevnar 13™; Test type: Other; p = 0.538, Miettinen & Nurminen; Difference in Percentage = 1.3, 95% CI 2-sided [-3.3 to 4.8] — V114 Combined Lots minus Prevnar 13™
Statistical Analysis 2: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Injection site pain: V114 Combined Lots - Prevnar 13™; Test type: Other; p < 0.001, Miettinen & Nurminen; Difference in Percentage = 14.6, 95% CI 2-sided [7.9 to 21.4] — V114 Combined Lots minus Prevnar 13™
Statistical Analysis 3: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Injection site swelling: V114 Combined Lots - Prevnar 13™; Test type: Other; p = 0.686, Miettinen & Nurminen; Difference in Percentage = 1.0, 95% CI 2-sided [-4.3 to 5.3] — V114 Combined Lots minus Prevnar 13™

3. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event Following Vaccination With Separate V114 Lots
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs consisted of muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue. The 95% CI were based on the exact binomial method proposed by Clopper and Pearson. Following vaccination with the three lots of V114 the percentage of participants with solicited systemic AEs was assessed. Per the statistical analysis plan, the Prevnar 13™ treatment group was not included as it was not analyzed with the same approach as the separate V114 lots.
Time Frame: Up to Day 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 699 | 704 | 700 | 0
Percentage of participants
  Arthralgia | 7.6 [5.7 to 9.8] | 7.0 [5.2 to 9.1] | 8.4 [6.5 to 10.7] |
  Fatigue | 22.0 [19.0 to 25.3] | 20.9 [17.9 to 24.1] | 21.6 [18.6 to 24.8] |
  Headache | 18.2 [15.4 to 21.2] | 19.9 [17.0 to 23.0] | 18.6 [15.8 to 21.7] |
  Myalgia | 28.0 [24.7 to 31.5] | 24.3 [21.2 to 27.6] | 28.4 [25.1 to 31.9] |

4. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event Following Vaccination: Combined Lots of V114 or Prevnar 13™
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs consisted of muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue. Per the statistical analysis plan, within-group CIs were not calculated.
Time Frame: Up to Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | V114 Combined Lots 1,2 and 3 | Prevnar13™
Number analyzed (Participants) | 2103 | 230
Percentage of participants
  Arthralgia | 7.7 | 5.7
  Fatigue | 21.5 | 22.2
  Headache | 18.9 | 18.7
  Myalgia | 26.9 | 21.7
Statistical Analysis 1: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Arthralgia: V114 Combined Lots - Prevnar 13™; Test type: Other; p = 0.272, Miettinen & Nurminen; Difference in Percentage = 2.0, 95% CI 2-sided [-1.9 to 4.7] — V114 Combined Lots minus Prevnar 13™
Statistical Analysis 2: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Fatigue: V114 Combined Lots - Prevnar 13™; Test type: Other; p = 0.812, Miettinen & Nurminen; Difference in Percentage = -0.7, 95% CI 2-sided [-6.7 to 4.5] — V114 Combined Lots minus Prevnar 13™
Statistical Analysis 3: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Headache: V114 Combined Lots - Prevnar 13™; Test type: Other; p = 0.947, Miettinen & Nurminen; Difference in Percentage = 0.2, 95% CI 2-sided [-5.6 to 5.0] — V114 Combined Lots minus Prevnar 13™
Statistical Analysis 4: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Myalgia: V114 Combined Lots - Prevnar 13™; Test type: Other; p = 0.091, Miettinen & Nurminen; Difference in Percentage = 5.2, 95% CI 2-sided [-0.9 to 10.4] — V114 Combined Lots minus Prevnar 13™

5. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event Following Vaccination With Separate V114 Lots
Description: A serious adverse event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. Relatedness of an SAE to the study vaccine is determined by the investigator. The 95% CI were based on the exact binomial method proposed by Clopper and Pearson. Following vaccination with the three lots of V114 the percentage of participants with SAEs was assessed. Per the statistical analysis plan, the Prevnar 13™ treatment group was not included as it was not analyzed with the same approach as the separate V114 lots.
Time Frame: Up to Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 699 | 704 | 700 | 0
Percentage of participants | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4] |

6. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event Following Vaccination: Combined Lots of V114 or Prevnar 13™
Description: A serious adverse event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. Relatedness of an SAE to the study vaccine is determined by the investigator. Per the statistical analysis plan, within-group CIs were not calculated.
Time Frame: Up to Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | V114 Combined Lots 1,2 and 3 | Prevnar13™
Number analyzed (Participants) | 2103 | 230
Percentage of participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; V114 Combined Lots - Prevnar 13™; Test type: Other; Miettinen & Nurminen = 0.0, 95% CI 2-sided [-1.6 to 0.2] — V114 Combined Lots minus Prevnar 13™

7. Primary Outcome: Geometric Mean Titer of Serotype-specific Opsonophagocytic Activity (OPA) Following Vaccination With Separate V114 Lots
Description: Opsonization of pneumococci for phagocytosis is an important mechanism by which antibodies to polysaccharides protect against disease in vivo. Sera from participants was used to measure geometric mean titer (GMT) of 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, using the Multiplexed Opsonophagocytic Assay (MOPA). Per the statistical analysis plan, within-group CIs were not calculated. 95% CIs were calculated for the GMT ratios between pairs of V114 lots by a constrained longitudinal data analysis (cLDA) model; and the Prevnar 13™ treatment group was not included as it was not analyzed with the same approach as the separate V114 lots.
Time Frame: Day 30
Population: All randomized participants without deviations from the protocol that may substantially affect the results of the outcome measure. Deviations include randomized but not vaccinated, missing results for serotypes, blood drawn out of time window, prohibited concomitant medication or vaccination.
Measure: Number; unit: 1/dil
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 698 | 704 | 700 | 0
1/dil
  Serotype 1: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 1 | 248.5 | 251.6 | 239.4 |
  Serotype 3: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 3 | 198.3 | 232.2 | 214.4 |
  Serotype 4: number analyzed (Participants) | 693 | 692 | 688 | 0
  Serotype 4 | 1073.1 | 1303.7 | 1074.4 |
  Serotype 5: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 5 | 389.8 | 461.6 | 391.3 |
  Serotype 6A: number analyzed (Participants) | 686 | 691 | 686 | 0
  Serotype 6A | 5845.0 | 6077.6 | 6123.8 |
  Serotype 6B: number analyzed (Participants) | 693 | 692 | 688 | 0
  Serotype 6B | 5160.6 | 5362.7 | 5109.5 |
  Serotype 7F: number analyzed (Participants) | 692 | 692 | 687 | 0
  Serotype 7F | 3757.7 | 4590.5 | 4202.0 |
  Serotype 9V: number analyzed (Participants) | 691 | 693 | 688 | 0
  Serotype 9V | 1708.4 | 1690.6 | 1749.9 |
  Serotype 14: number analyzed (Participants) | 693 | 693 | 687 | 0
  Serotype 14 | 2364.8 | 2509.6 | 2050.6 |
  Serotype 18C: number analyzed (Participants) | 693 | 692 | 688 | 0
  Serotype 18C | 3880.8 | 3522.4 | 3381.0 |
  Serotype 19A: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 19A | 3384.7 | 3774.8 | 3498.5 |
  Serotype 19F: number analyzed (Participants) | 693 | 692 | 688 | 0
  Serotype 19F | 1866.4 | 2017.8 | 1993.2 |
  Serotype 23F: number analyzed (Participants) | 690 | 692 | 686 | 0
  Serotype 23F | 2222.9 | 2417.8 | 2133.0 |
  Serotype 22F: number analyzed (Participants) | 688 | 692 | 684 | 0
  Serotype 22F | 2617.4 | 2761.6 | 2676.0 |
  Serotype 33F: number analyzed (Participants) | 691 | 690 | 688 | 0
  Serotype 33F | 7758.1 | 7736.9 | 7365.6 |
Statistical Analysis 1: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 1: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; P-value for the comparison of the GMT ratio to the lower bound (0.5). P-value for the comparison of the GMT ratio to the upper bound (2.0); GMT Ratio = 0.99, 95% CI 2-sided [0.83 to 1.18] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 2: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 1: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.04, 95% CI 2-sided [0.87 to 1.24] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 3: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 1: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.05, 95% CI 2-sided [0.88 to 1.25] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 4: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 3: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.85, 95% CI 2-sided [0.75 to 0.97] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 5: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 3: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.92, 95% CI 2-sided [0.81 to 1.05] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 6: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 3: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.08, 95% CI 2-sided [0.95 to 1.23] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 7: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 4: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.82, 95% CI 2-sided [0.70 to 0.97] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 8: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 4: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.85 to 1.18] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 9: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 4: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.21, 95% CI 2-sided [1.03 to 1.43] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 10: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 5: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.84, 95% CI 2-sided [0.70 to 1.02] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 11: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 5: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.83 to 1.20] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 12: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 5: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.18, 95% CI 2-sided [0.98 to 1.42] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 13: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 6A: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.96, 95% CI 2-sided [0.82 to 1.12] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 14: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 6A: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.95, 95% CI 2-sided [0.82 to 1.12] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 15: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 6A: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.99, 95% CI 2-sided [0.85 to 1.16] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 16: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 6B: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.96, 95% CI 2-sided [0.82 to 1.12] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 17: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 6B: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.01, 95% CI 2-sided [0.86 to 1.18] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 18: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 6B: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.05, 95% CI 2-sided [0.90 to 1.23] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 19: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 7F: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.82, 95% CI 2-sided [0.72 to 0.93] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 20: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 7F: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.89, 95% CI 2-sided [0.79 to 1.01] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 21: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 7F: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.09, 95% CI 2-sided [0.96 to 1.24] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 22: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 9V: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.01, 95% CI 2-sided [0.88 to 1.16] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 23: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 9V: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.98, 95% CI 2-sided [0.85 to 1.12] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 24: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 9V: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.97, 95% CI 2-sided [0.84 to 1.11] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 25: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 14: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.94, 95% CI 2-sided [0.81 to 1.10] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 26: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 14: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.15, 95% CI 2-sided [0.99 to 1.34] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 27: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 14: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.22, 95% CI 2-sided [1.05 to 1.43] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 28: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 18C: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.10, 95% CI 2-sided [0.96 to 1.26] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 29: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 18C: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.15, 95% CI 2-sided [1.00 to 1.31] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 30: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 18C: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.04, 95% CI 2-sided [0.91 to 1.19] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 31: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 19A: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.90, 95% CI 2-sided [0.79 to 1.02] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 32: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 19A: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.97, 95% CI 2-sided [0.85 to 1.10] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 33: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 19A: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.08, 95% CI 2-sided [0.95 to 1.22] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 34: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 19F: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.92, 95% CI 2-sided [0.81 to 1.05] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 35: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 19F: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.94, 95% CI 2-sided [0.82 to 1.07] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 36: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 19F: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.01, 95% CI 2-sided [0.89 to 1.15] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 37: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 23F: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.92, 95% CI 2-sided [0.77 to 1.10] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 38: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 23F: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.04, 95% CI 2-sided [0.87 to 1.24] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 39: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 23F: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.13, 95% CI 2-sided [0.95 to 1.35] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 40: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 22F: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.95, 95% CI 2-sided [0.81 to 1.11] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 41: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 22F: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.98, 95% CI 2-sided [0.84 to 1.14] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 42: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 22F: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.03, 95% CI 2-sided [0.88 to 1.21] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 43: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 33F: GMT Ratio V114 Lot 1 / V114 Lot 2; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.86 to 1.16] — Lot 1 divided by Lot 2; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 44: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 33F: GMT Ratio V114 Lot 1 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.05, 95% CI 2-sided [0.91 to 1.22] — Lot 1 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 45: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 33F: GMT Ratio V114 Lot 2 / V114 Lot 3; Test type: Equivalence — Lower and upper p-values ≤ 0.025 support a conclusion of equivalence; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.05, 95% CI 2-sided [0.90 to 1.22] — Lot 2 divided by Lot 3; GMT ratio and 95% CI were estimated from a cLDA model

8. Secondary Outcome: Geometric Mean Concentration of Serotype-specific Immunoglobulin G (IgG) Following Vaccination With Separate V114 Lots
Description: The geometric mean concentration (GMC) of IgG serotype-specific antibodies to the 13 pneumococcal polysaccharide serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) contained in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, were quantitated from participants' sera by multiplex electrochemiluminescence (ECL) using the pneumococcal electrochemiluminescence (PnECL) v2.0 assay. Per the statistical analysis plan, within-group CIs were not calculated; and the Prevnar 13™ treatment group was not included as it was not analyzed with the same approach as the separate V114 lots.
Time Frame: Day 30
Population: as for outcome 7
Measure: Number; unit: μg/mL
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 698 | 704 | 700 | 0
μg/mL
  Serotype 1: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 1 | 3.91 | 4.05 | 3.83 |
  Serotype 3: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 3 | 0.74 | 0.86 | 0.73 |
  Serotype 4: number analyzed (Participants) | 693 | 692 | 688 | 0
  Serotype 4 | 1.79 | 2.18 | 1.67 |
  Serotype 5: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 5 | 3.81 | 4.63 | 3.96 |
  Serotype 6A: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 6A | 8.09 | 8.84 | 8.16 |
  Serotype 6B: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 6B | 10.92 | 11.46 | 10.44 |
  Serotype 7F: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 7F | 5.71 | 7.11 | 5.94 |
  Serotype 9V: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 9V | 4.20 | 4.44 | 4.26 |
  Serotype 14: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 14 | 9.82 | 11.38 | 8.66 |
  Serotype 18C: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 18C | 14.07 | 11.81 | 10.66 |
  Serotype 19A: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 19A | 15.45 | 17.34 | 15.81 |
  Serotype 19F: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 19F | 9.78 | 11.22 | 10.65 |
  Serotype 23F: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 23F | 7.38 | 7.97 | 7.44 |
  Serotype 22F: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 22F | 4.12 | 4.41 | 3.80 |
  Serotype 33F: number analyzed (Participants) | 693 | 693 | 688 | 0
  Serotype 33F | 9.92 | 10.88 | 9.45 |
Statistical Analysis 1: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 1: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.96, 95% CI 2-sided [0.84 to 1.10] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 2: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 1: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 1.02, 95% CI 2-sided [0.89 to 1.17] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 3: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 1: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.06, 95% CI 2-sided [0.92 to 1.21] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 4: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 3: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.85, 95% CI 2-sided [0.77 to 0.95] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 5: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 3: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.91 to 1.13] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 6: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 3: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.18, 95% CI 2-sided [1.06 to 1.32] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 7: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 4: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.82, 95% CI 2-sided [0.72 to 0.94] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 8: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 4: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 1.07, 95% CI 2-sided [0.94 to 1.23] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 9: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 4: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; P-value for the comparison of the GMT ratio to the upper bound (2.0); GMC Ratio = 1.31, 95% CI 2-sided [1.14 to 1.50] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 10: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 5: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.82, 95% CI 2-sided [0.72 to 0.95] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 11: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 5: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 0.96, 95% CI 2-sided [0.84 to 1.11] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 12: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 5: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.17, 95% CI 2-sided [1.02 to 1.35] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 13: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 6A: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.92, 95% CI 2-sided [0.78 to 1.07] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 14: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 6A: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.85 to 1.16] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 15: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 6A: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.08, 95% CI 2-sided [0.93 to 1.27] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 16: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 6B: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.95, 95% CI 2-sided [0.82 to 1.11] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 17: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 6B: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 1.05, 95% CI 2-sided [0.90 to 1.22] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 18: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 6B: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.10, 95% CI 2-sided [0.94 to 1.28] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 19: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 7F: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.80, 95% CI 2-sided [0.70 to 0.92] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 20: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 7F: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 0.96, 95% CI 2-sided [0.84 to 1.10] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 21: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 7F: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.20, 95% CI 2-sided [1.04 to 1.37] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 22: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 9V: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; l; GMC Ratio = 0.95, 95% CI 2-sided [0.83 to 1.08] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 23: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 9V: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.87 to 1.13] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 24: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 9V: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.04, 95% CI 2-sided [0.91 to 1.19] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 25: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 14: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.86, 95% CI 2-sided [0.75 to 1.00] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 26: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 14: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 1.13, 95% CI 2-sided [0.98 to 1.31] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 27: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 14: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.31, 95% CI 2-sided [1.14 to 1.52] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 28: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 18C: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 1.19, 95% CI 2-sided [1.04 to 1.36] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 29: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 18C: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 1.32, 95% CI 2-sided [1.15 to 1.51] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 30: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 18C: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.11, 95% CI 2-sided [0.97 to 1.27] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 31: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 19A: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.89, 95% CI 2-sided [0.78 to 1.02] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 32: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 19A: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 0.98, 95% CI 2-sided [0.86 to 1.11] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 33: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 19A: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.10, 95% CI 2-sided [0.96 to 1.25] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 34: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 19F: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.87, 95% CI 2-sided [0.76 to 1.00] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 35: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 19F: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 0.92, 95% CI 2-sided [0.80 to 1.05] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 36: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 19F: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.05, 95% CI 2-sided [0.92 to 1.21] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 37: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 23F: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.93, 95% CI 2-sided [0.80 to 1.07] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 38: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 23F: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.86 to 1.15] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 39: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 23F: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.07, 95% CI 2-sided [0.93 to 1.24] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 40: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 22F: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.93, 95% CI 2-sided [0.81 to 1.08] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 41: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 22F: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 1.08, 95% CI 2-sided [0.93 to 1.26] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 42: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 22F: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.16, 95% CI 2-sided [1.00 to 1.35] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 43: Comparison: V114 Lot 1 vs V114 Lot 2; Serotype 33F: GMC Ratio V114 Lot 1 / V114 Lot 2; Test type: Other; GMC Ratio = 0.91, 95% CI 2-sided [0.79 to 1.06] — Lot 1 divided by Lot 2; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 44: Comparison: V114 Lot 1 vs V114 Lot 3; Serotype 33F: GMC Ratio V114 Lot 1 / V114 Lot 3; Test type: Other; GMC Ratio = 1.05, 95% CI 2-sided [0.90 to 1.22] — Lot 1 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 45: Comparison: V114 Lot 2 vs V114 Lot 3; Serotype 33F: GMC Ratio V114 Lot 2 / V114 Lot 3; Test type: Other; GMC Ratio = 1.15, 95% CI 2-sided [0.99 to 1.34] — Lot 2 divided by Lot 3; GMC ratio and 95% CI were estimated from a cLDA model

9. Secondary Outcome: Geometric Mean Concentration of Serotype-specific IgG Following Vaccination: Combined Lots of V114 or Prevnar 13™
Description: The GMC of IgG serotype-specific antibodies to the 13 pneumococcal polysaccharide serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) contained in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, were quantitated from participants' sera by ECL. Per the statistical analysis plan, within-group CIs were not calculated,
Time Frame: Day 30
Population: as for outcome 7
Measure: Number; unit: μg/mL
Arm/Group | V114 Combined Lots 1,2 and 3 | Prevnar13™
Number analyzed (Participants) | 2102 | 231
μg/mL
  Serotype 1: number analyzed (Participants) | 2074 | 225
  Serotype 1 | 3.91 | 5.22
  Serotype 3: number analyzed (Participants) | 2074 | 225
  Serotype 3 | 0.77 | 0.55
  Serotype 4: number analyzed (Participants) | 2073 | 225
  Serotype 4 | 1.87 | 2.38
  Serotype 5: number analyzed (Participants) | 2074 | 225
  Serotype 5 | 4.14 | 4.66
  Serotype 6A: number analyzed (Participants) | 2074 | 225
  Serotype 6A | 8.38 | 7.20
  Serotype 6B: number analyzed (Participants) | 2074 | 225
  Serotype 6B | 10.92 | 7.28
  Serotype 7F: number analyzed (Participants) | 2074 | 225
  Serotype 7F | 6.19 | 7.12
  Serotype 9V: number analyzed (Participants) | 2074 | 225
  Serotype 9V | 4.30 | 4.97
  Serotype 14: number analyzed (Participants) | 2074 | 225
  Serotype 14 | 9.89 | 9.97
  Serotype 18C: number analyzed (Participants) | 2074 | 225
  Serotype 18C | 12.08 | 9.58
  Serotype 19A: number analyzed (Participants) | 2074 | 225
  Serotype 19A | 16.18 | 16.66
  Serotype 19F: number analyzed (Participants) | 2074 | 225
  Serotype 19F | 10.52 | 10.25
  Serotype 23F: number analyzed (Participants) | 2074 | 225
  Serotype 23F | 7.58 | 6.03
  Serotype 22F: number analyzed (Participants) | 2074 | 225
  Serotype 22F | 4.10 | 0.34
  Serotype 33F: number analyzed (Participants) | 2074 | 225
  Serotype 33F | 10.03 | 1.07
Statistical Analysis 1: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 1: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 0.75, 95% CI 2-sided [0.62 to 0.91] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 2: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 3: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 1.39, 95% CI 2-sided [1.20 to 1.61] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 3: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 4: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 0.79, 95% CI 2-sided [0.66 to 0.94] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 4: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 5: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 0.89, 95% CI 2-sided [0.74 to 1.07] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 5: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 6A: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 1.16, 95% CI 2-sided [0.95 to 1.43] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 6: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 6B: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 1.50, 95% CI 2-sided [1.21 to 1.86] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 7: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 7F: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 0.87, 95% CI 2-sided [0.73 to 1.04] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 8: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 9V: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 0.87, 95% CI 2-sided [0.72 to 1.04] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 9: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 14: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.82 to 1.20] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 10: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 18C: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 1.26, 95% CI 2-sided [1.05 to 1.51] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 11: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 19A: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 0.97, 95% CI 2-sided [0.82 to 1.15] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 12: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 19F: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 1.03, 95% CI 2-sided [0.86 to 1.23] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 13: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 23F: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 1.26, 95% CI 2-sided [1.03 to 1.54] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 14: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 22F: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 12.21, 95% CI 2-sided [10.11 to 14.74] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 15: Comparison: V114 Combined Lots 1,2 and 3 vs Prevnar13™; Serotype 33F: GMC Ratio V114 Combined Lots / Prevnar 13™; Test type: Other; GMC Ratio = 9.42, 95% CI 2-sided [7.96 to 11.13] — V114 Combined Lots divided by Prevnar 13™; GMC ratio and 95% CI were estimated from a cLDA model

10. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Serotype-specific OPA Following Vaccination With Separate V114 Lots
Description: Sera from participants was used to measure GMT of 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, using the MOPA which reads the reciprocal of the highest dilution that gives ≥50% bacterial killing. The Geometric Mean Fold Rise (GMFR) is the geometric mean of the ratio Day 30/Day 1 OPA responses. Per the statistical analysis plan, the Prevnar 13™ treatment group was not analyzed.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 698 | 704 | 700 | 0
Ratio
  Serotype 1: number analyzed (Participants) | 676 | 667 | 661 | 0
  Serotype 1 | 15.9 [13.9 to 18.2] | 16.5 [14.6 to 18.8] | 15.4 [13.6 to 17.4] |
  Serotype 3: number analyzed (Participants) | 666 | 665 | 657 | 0
  Serotype 3 | 6.5 [5.9 to 7.2] | 7.6 [6.8 to 8.4] | 6.9 [6.2 to 7.6] |
  Serotype 4: number analyzed (Participants) | 670 | 663 | 658 | 0
  Serotype 4 | 17.4 [15.4 to 19.8] | 20.7 [18.3 to 23.4] | 16.5 [14.6 to 18.7] |
  Serotype 5: number analyzed (Participants) | 676 | 675 | 665 | 0
  Serotype 5 | 11.2 [9.9 to 12.8] | 13.3 [11.8 to 15.1] | 11.1 [9.8 to 12.7] |
  Serotype 6A: number analyzed (Participants) | 620 | 618 | 611 | 0
  Serotype 6A | 13.7 [12.1 to 15.5] | 14.1 [12.5 to 16.0] | 14.6 [12.8 to 16.5] |
  Serotype 6B: number analyzed (Participants) | 659 | 658 | 653 | 0
  Serotype 6B | 33.4 [29.0 to 38.5] | 31.2 [27.0 to 36.1] | 34.9 [30.2 to 40.3] |
  Serotype 7F: number analyzed (Participants) | 648 | 638 | 646 | 0
  Serotype 7F | 11.9 [10.4 to 13.7] | 14.3 [12.4 to 16.5] | 12.9 [11.3 to 14.8] |
  Serotype 9V: number analyzed (Participants) | 652 | 650 | 641 | 0
  Serotype 9V | 4.8 [4.4 to 5.3] | 4.8 [4.3 to 5.3] | 5.0 [4.5 to 5.6] |
  Serotype 14: number analyzed (Participants) | 671 | 667 | 662 | 0
  Serotype 14 | 7.6 [6.6 to 8.6] | 7.6 [6.7 to 8.7] | 6.2 [5.4 to 7.0] |
  Serotype 18C: number analyzed (Participants) | 669 | 662 | 651 | 0
  Serotype 18C | 16.7 [14.9 to 18.8] | 15.0 [13.4 to 16.8] | 14.1 [12.6 to 15.8] |
  Serotype 19A: number analyzed (Participants) | 665 | 660 | 650 | 0
  Serotype 19A | 10.4 [9.2 to 11.8] | 11.0 [9.6 to 12.5] | 11.7 [10.3 to 13.4] |
  Serotype 19F: number analyzed (Participants) | 663 | 667 | 659 | 0
  Serotype 19F | 6.5 [5.9 to 7.3] | 6.8 [6.1 to 7.6] | 7.3 [6.5 to 8.1] |
  Serotype 23F: number analyzed (Participants) | 609 | 626 | 633 | 0
  Serotype 23F | 16.8 [14.6 to 19.4] | 17.4 [15.2 to 20.0] | 17.0 [14.8 to 19.4] |
  Serotype 22F: number analyzed (Participants) | 610 | 597 | 602 | 0
  Serotype 22F | 27.2 [22.3 to 33.1] | 31.1 [25.6 to 38.0] | 28.3 [23.4 to 34.3] |
  Serotype 33F: number analyzed (Participants) | 647 | 641 | 641 | 0
  Serotype 33F | 8.4 [7.2 to 9.7] | 7.7 [6.6 to 8.9] | 7.5 [6.5 to 8.7] |

11. Secondary Outcome: GMFR in Serotype-specific IgG Following Vaccination With Separate V114 Lots
Description: The geometric mean concentration (GMC) of IgG serotype-specific antibodies to the 13 pneumococcal polysaccharide serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) contained in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, were quantitated from participants' sera by ECL. The GMFR is the geometric mean of the ratio Day 30/Day 1 IgG concentration. Per the statistical analysis plan, the Prevnar 13™ treatment group was not analyzed.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 698 | 704 | 700 | 0
Ratio
  Serotype 1: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 1 | 10.9 [9.8 to 12.2] | 11.2 [10.1 to 12.4] | 10.3 [9.2 to 11.5] |
  Serotype 3: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 3 | 5.4 [4.9 to 5.9] | 6.3 [5.7 to 6.9] | 5.2 [4.8 to 5.7] |
  Serotype 4: number analyzed (Participants) | 673 | 672 | 664 | 0
  Serotype 4 | 8.6 [7.8 to 9.5] | 10.5 [9.5 to 11.6] | 7.9 [7.1 to 8.7] |
  Serotype 5: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 5 | 4.5 [4.1 to 5.0] | 5.5 [4.9 to 6.0] | 4.7 [4.2 to 5.2] |
  Serotype 6A: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 6A | 22.6 [20.1 to 25.3] | 24.1 [21.5 to 27.1] | 22.9 [20.4 to 25.8] |
  Serotype 6B: number analyzed (Participants) | 676 | 674 | 666 | 0
  Serotype 6B | 23.5 [21.0 to 26.3] | 24.1 [21.5 to 27.0] | 22.1 [19.7 to 24.8] |
  Serotype 7F: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 7F | 11.7 [10.5 to 13.1] | 14.8 [13.2 to 16.6] | 12.0 [10.7 to 13.3] |
  Serotype 9V: number analyzed (Participants) | 676 | 673 | 665 | 0
  Serotype 9V | 9.5 [8.6 to 10.5] | 9.8 [8.9 to 10.9] | 9.6 [8.6 to 10.6] |
  Serotype 14: number analyzed (Participants) | 676 | 674 | 666 | 0
  Serotype 14 | 6.5 [5.8 to 7.3] | 6.8 [6.1 to 7.7] | 5.2 [4.7 to 5.8] |
  Serotype 18C: number analyzed (Participants) | 676 | 674 | 666 | 0
  Serotype 18C | 20.6 [18.3 to 23.1] | 17.0 [15.1 to 19.1] | 15.9 [14.2 to 17.9] |
  Serotype 19A: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 19A | 9.1 [8.2 to 10.0] | 10.6 [9.6 to 11.7] | 9.5 [8.6 to 10.5] |
  Serotype 19F: number analyzed (Participants) | 677 | 673 | 665 | 0
  Serotype 19F | 12.3 [11.1 to 13.7] | 13.8 [12.5 to 15.4] | 13.1 [11.8 to 14.5] |
  Serotype 23F: number analyzed (Participants) | 677 | 674 | 665 | 0
  Serotype 23F | 14.3 [12.7 to 16.1] | 16.2 [14.4 to 18.1] | 14.8 [13.2 to 16.6] |
  Serotype 22F: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 22F | 12.8 [11.4 to 14.4] | 13.4 [11.8 to 15.1] | 11.1 [9.9 to 12.5] |
  Serotype 33F: number analyzed (Participants) | 677 | 673 | 666 | 0
  Serotype 33F | 9.2 [8.3 to 10.3] | 9.5 [8.6 to 10.6] | 7.9 [7.1 to 8.8] |

12. Secondary Outcome: Percentage of Participants With ≥4 Fold Change in Serotype-specific OPA Following Vaccination With Separate V114 Lots
Description: Sera from participants was used to measure GMT of 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, with the MOPA which reads the reciprocal of the highest dilution (1/dil) that gives ≥50% bacterial killing. Percentage of participants with a ≥ 4-fold change from Day 1 (baseline) to Day 30 (Day 30/Day 1) are presented. Per the statistical analysis plan, the Prevnar 13™ treatment group was not analyzed.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 698 | 704 | 700 | 0
Percentage of participants
  Serotype 1: number analyzed (Participants) | 676 | 667 | 661 | 0
  Serotype 1 | 74.4 [70.9 to 77.7] | 76.8 [73.4 to 79.9] | 77.2 [73.8 to 80.3] |
  Serotype 3: number analyzed (Participants) | 666 | 665 | 657 | 0
  Serotype 3 | 64.7 [61.0 to 68.3] | 68.9 [65.2 to 72.4] | 64.8 [61.1 to 68.5] |
  Serotype 4: number analyzed (Participants) | 670 | 663 | 658 | 0
  Serotype 4 | 79.4 [76.1 to 82.4] | 83.6 [80.5 to 86.3] | 79.5 [76.2 to 82.5] |
  Serotype 5: number analyzed (Participants) | 676 | 675 | 665 | 0
  Serotype 5 | 71.3 [67.7 to 74.7] | 76.1 [72.7 to 79.3] | 69.5 [65.8 to 73.0] |
  Serotype 6A: number analyzed (Participants) | 620 | 618 | 611 | 0
  Serotype 6A | 78.5 [75.1 to 81.7] | 77.8 [74.3 to 81.0] | 76.9 [73.4 to 80.2] |
  Serotype 6B: number analyzed (Participants) | 659 | 658 | 653 | 0
  Serotype 6B | 83.3 [80.2 to 86.1] | 83.6 [80.5 to 86.3] | 84.5 [81.5 to 87.2] |
  Serotype 7F: number analyzed (Participants) | 648 | 638 | 646 | 0
  Serotype 7F | 69.4 [65.7 to 73.0] | 71.6 [68.0 to 75.1] | 70.4 [66.7 to 73.9] |
  Serotype 9V: number analyzed (Participants) | 652 | 650 | 641 | 0
  Serotype 9V | 53.4 [49.5 to 57.3] | 51.2 [47.3 to 55.1] | 53.2 [49.3 to 57.1] |
  Serotype 14: number analyzed (Participants) | 671 | 667 | 662 | 0
  Serotype 14 | 56.8 [52.9 to 60.6] | 57.6 [53.7 to 61.4] | 52.3 [48.4 to 56.1] |
  Serotype 18C: number analyzed (Participants) | 669 | 662 | 651 | 0
  Serotype 18C | 80.1 [76.9 to 83.1] | 79.0 [75.7 to 82.0] | 78.3 [75.0 to 81.4] |
  Serotype 19A: number analyzed (Participants) | 665 | 660 | 650 | 0
  Serotype 19A | 67.8 [64.1 to 71.4] | 69.8 [66.2 to 73.3] | 71.2 [67.6 to 74.7] |
  Serotype 19F: number analyzed (Participants) | 663 | 667 | 659 | 0
  Serotype 19F | 60.8 [57.0 to 64.5] | 61.9 [58.1 to 65.6] | 63.0 [59.2 to 66.7] |
  Serotype 23F: number analyzed (Participants) | 609 | 626 | 633 | 0
  Serotype 23F | 75.4 [71.7 to 78.7] | 78.3 [74.8 to 81.4] | 78.2 [74.8 to 81.4] |
  Serotype 22F: number analyzed (Participants) | 610 | 597 | 602 | 0
  Serotype 22F | 71.1 [67.4 to 74.7] | 73.4 [69.6 to 76.9] | 72.8 [69.0 to 76.3] |
  Serotype 33F: number analyzed (Participants) | 647 | 641 | 641 | 0
  Serotype 33F | 59.5 [55.6 to 63.3] | 58.3 [54.4 to 62.2] | 56.8 [52.8 to 60.7] |

13. Secondary Outcome: Percentage of Participants With ≥4 Fold Change in Serotype-specific IgG Following Vaccination With Separate V114 Lots
Description: The geometric mean concentration of IgG serotype-specific antibodies to the 13 pneumococcal polysaccharide serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) contained in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, were quantitated from participants' sera by ECL. Percentage of participants with a ≥ 4-fold change from Day 1 (baseline) to Day 30 (Day 30/ Day 1) are presented. Per the statistical analysis plan, the Prevnar 13™ treatment group was not analyzed.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar13™
Number analyzed (Participants) | 698 | 704 | 700 | 0
Percentage of participants
  Serotype 1: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 1 | 73.9 [70.4 to 77.1] | 75.2 [71.8 to 78.4] | 73.0 [69.4 to 76.3] |
  Serotype 3: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 3 | 58.6 [54.8 to 62.4] | 61.9 [58.1 to 65.6] | 54.7 [50.8 to 58.5] |
  Serotype 4: number analyzed (Participants) | 673 | 672 | 664 | 0
  Serotype 4 | 68.8 [65.1 to 72.3] | 73.8 [70.3 to 77.1] | 65.7 [61.9 to 69.3] |
  Serotype 5: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 5 | 45.6 [41.8 to 49.5] | 52.5 [48.7 to 56.3] | 45.9 [42.1 to 49.8] |
  Serotype 6A: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 6A | 86.6 [83.8 to 89.0] | 87.2 [84.5 to 89.7] | 83.8 [80.8 to 86.5] |
  Serotype 6B: number analyzed (Participants) | 676 | 674 | 666 | 0
  Serotype 6B | 87.0 [84.2 to 89.4] | 85.6 [82.7 to 88.2] | 84.2 [81.2 to 86.9] |
  Serotype 7F: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 7F | 75.3 [71.9 to 78.5] | 78.8 [75.5 to 81.8] | 74.8 [71.3 to 78.0] |
  Serotype 9V: number analyzed (Participants) | 676 | 673 | 665 | 0
  Serotype 9V | 72.6 [69.1 to 76.0] | 73.0 [69.4 to 76.3] | 71.6 [68.0 to 75.0] |
  Serotype 14: number analyzed (Participants) | 676 | 674 | 666 | 0
  Serotype 14 | 54.4 [50.6 to 58.2] | 57.9 [54.0 to 61.6] | 48.3 [44.5 to 52.2] |
  Serotype 18C: number analyzed (Participants) | 676 | 674 | 666 | 0
  Serotype 18C | 84.6 [81.7 to 87.3] | 78.6 [75.3 to 81.7] | 76.7 [73.3 to 79.9] |
  Serotype 19A: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 19A | 70.6 [67.0 to 74.0] | 74.2 [70.7 to 77.5] | 71.0 [67.4 to 74.4] |
  Serotype 19F: number analyzed (Participants) | 677 | 673 | 665 | 0
  Serotype 19F | 77.8 [74.5 to 80.9] | 79.0 [75.8 to 82.1] | 78.6 [75.3 to 81.7] |
  Serotype 23F: number analyzed (Participants) | 677 | 674 | 665 | 0
  Serotype 23F | 76.1 [72.7 to 79.2] | 80.7 [77.5 to 83.6] | 76.7 [73.3 to 79.9] |
  Serotype 22F: number analyzed (Participants) | 677 | 674 | 666 | 0
  Serotype 22F | 75.3 [71.9 to 78.5] | 75.4 [71.9 to 78.6] | 72.1 [68.5 to 75.5] |
  Serotype 33F: number analyzed (Participants) | 677 | 673 | 666 | 0
  Serotype 33F | 69.4 [65.8 to 72.9] | 70.9 [67.3 to 74.3] | 66.1 [62.3 to 69.7] |

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs) were reported from Day 1 through Day 14 following vaccination. Serious AEs (SAEs) were reported from Day 1 following vaccination up to Month 6. All-Cause Mortality were reported from randomization up to Month 6.
Description: For SAEs and Non-serious AEs the population analyzed was randomized participants according to the intervention they actually received. One participant randomized to the Prevnar 13™ group incorrectly received V114 Lot 1. For All-Cause Mortality the population analyzed was all randomized participants.
Arm/Group | V114 Lot 1 | V114 Lot 2 | V114 Lot 3 | Prevnar 13™
All-Cause Mortality (participants affected / at risk) | 1/702 | 2/704 | 0/701 | 0/233
Serious Adverse Events (participants affected / at risk) | 12/699 | 19/704 | 7/700 | 5/230
Other Adverse Events (participants affected / at risk) | 548/699 | 534/704 | 535/700 | 151/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 Lot 1 (N=699) | V114 Lot 2 (N=704) | V114 Lot 3 (N=700) | Prevnar 13™ (N=230)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Due to unknown cause
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 Lot 1 (N=699) | V114 Lot 2 (N=704) | V114 Lot 3 (N=700) | Prevnar 13™ (N=230)
Fatigue (General disorders) | 154 (202) | 147 (182) | 151 (189) | 51 (74)
Injection site erythema (General disorders) | 77 (82) | 86 (91) | 89 (91) | 22 (24)
Injection site pain (General disorders) | 464 (518) | 475 (520) | 471 (514) | 122 (134)
Injection site swelling (General disorders) | 111 (115) | 115 (117) | 106 (109) | 34 (34)
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 (68) | 49 (54) | 59 (75) | 13 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 196 (226) | 171 (196) | 199 (226) | 50 (54)
Headache (Nervous system disorders) | 127 (166) | 140 (170) | 130 (171) | 43 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT03950856/Prot_SAP_000.pdf